CLINICAL TRIAL: NCT04514679
Title: Randomize Everyone: Creating Valid Instrumental Variables for Learning Health Care Systems
Brief Title: EHR Embedded Comparative Effectiveness Studies--WWC
Acronym: EHR-WWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Trustees of Dartmouth College (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Tor D. Tosteson, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D19107a
Record Dates: First submitted 2020-01-10; First posted 2020-08-17 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietician / Health Coach (Active Comparator): Patients having obesity treatment would first see a dietician, and then see a health coach.
  Interventions: Behavioral: Dietician / Health Coach
- Health Coach / Dietician (Active Comparator): Patients having obesity treatment would first see a health coach, and then see a dietician.
  Interventions: Behavioral: Health Coach / Dietician

INTERVENTIONS:
Behavioral: Dietician / Health Coach — The order of visit for the two types of providers is first Dietician then Health Coach.
  Arms: Dietician / Health Coach
Behavioral: Health Coach / Dietician — The order of visit for the two types of providers is first Health Coach then Dietician.
  Arms: Health Coach / Dietician

SUMMARY:
Randomize Everyone is a research project to develop new informatics systems and statistical methods for supporting randomization processes in EHR systems to do comparative effectiveness research. Two demonstration projects are being conducted in the Dartmouth Hitchcock Medical Center, designed to evaluate different weight loss interventions and common practices in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
EHR Embedded Comparative Effectiveness Studies-WWC will be held in the Weight and Wellness Clinics at Dartmouth-Hitchcock Medical Center. This study consists of randomizing enrollees to either the dietitian/health coach appointment sequence or the health coach/dietitian appointment sequence.

ELIGIBILITY:
Inclusion Criteria: Adults (>18) able to consent, with sufficient fluency in English; Initial RD and HC visits are part of routine care as recommended by the provider; willing to be randomized

Exclusion Criteria: Pregnant women; Prisoners; Children (<18)

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dietician / Health Coach | Health Coach / Dietician
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age was unavailable due to missing data in the patient record.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietician / Health Coach | Health Coach / Dietician | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (14.4) | 45.2 (13.5) | 45.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Compliance Rate
Description: Percentage of those in each arm who complete the two visits in the correct order assigned.
Time Frame: Baseline through approximately 2 months
Population: Those who had health record data, which eliminated 3 patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dietician / Health Coach | Health Coach / Dietician
Number analyzed (Participants) | 28 | 29
percentage of participants | 87 [66 to 97] | 76 [54 to 90]

2. Primary Outcome: Percentage of Eligible Patients Participating
Description: Percentage of those identified as being eligible who were enrolled in the study.
Time Frame: One day, during the recruitment period of October 23, 2020 to February 3, 2021.
Population: All patients who were identified as being eligible.
Measure: Number (95% Confidence Interval); unit: percentage of eligible patients
Groups:
- All Eligible Patients: All eligible patients approached to participate.
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 459
percentage of eligible patients | 13.1 [10.2 to 16.6]

3. Secondary Outcome: Change in Body Mass Index (BMI) at 30 Days
Description: Linear trends (or "slopes") for per 30 days are calculated in each group. The slopes were calculated from repeated BMI measurements in each treatment group, and expressed in terms of the change in BMI predicted at 30 days post randomization.
Time Frame: 30 days since baseline
Population: Those who had health record data, which eliminated 3 patients.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Dietician / Health Coach | Health Coach / Dietician
Number analyzed (Participants) | 28 | 29
kg/m^2 | -0.07 (0.25) | -0.16 (0.20)

ADVERSE EVENTS:
Time Frame: 6 months post randomization
Description: Adverse events were assessed by the participating clinic as part of routine clinical practice.
Arm/Group | Dietician / Health Coach | Health Coach / Dietician
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This study is part of a project that evaluates the utility of methods to use randomized methods for evaluating comparative effectiveness questions using the electronic health record of a health system. The primary focus is on the feasibility of the method, including the patient participation and compliance rates for an intervention in an obesity clinic involving timing of visits to a health coach and a dietician. The results regarding the efficacy of the intervention are secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT04514679/Prot_SAP_000.pdf